CLINICAL TRIAL: NCT02881801
Title: Patterns of Physical Activity and Sedentary Time in Survivors of a Critical Illness During a Hospital Admission
Status: Completed | Type: Observational
Sponsor: University of South Australia (Other)
Collaborators: Australian Physiotherapy Research Foundation (Other); University of Leicester (Other)
Responsible Party: Principal Investigator, Claire Baldwin, Principal Investigator, University of South Australia
Other Study IDs: 0000032489; 91.41 (Other: Southern Adelaide Health Service)
Record Dates: First submitted 2016-08-03; First posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Motor Activity; Sedentary Lifestyle; Critical Illness
Keywords: accelerometry
MeSH Terms: conditions — Motor Activity; Sedentary Behavior; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to describe the pattern of active and sedentary time in survivors of a critical illness, at three time points during their hospital admission (awakening in the ICU after ≥ 5 days of mechanical ventilation, discharge to ward and discharge from hospital).

The specific research objectives are to

1. Determine the duration of active and sedentary parameters including time and bouts in 24 hour periods
2. Examine changes in the active and sedentary parameters including time and bouts between time points of awakening and both ICU and hospital discharge.
3. Conduct a preliminary examination of relationships between activity and sedentary behaviour metrics with measures of muscle strength, physical function and hospital length of stay.

DETAILED DESCRIPTION:
This is a prospective observational study that consecutively samples eligible patients with a critical illness, requiring intensive care. This study will use two activity monitors (accelerometers) to measure physical activity and sedentary variables from patients recovering from a critical illness in a single tertiary hospital on three occasions during their acute hospital admission. Accelerometer derived measures will be obtained from continuous 24 hour monitoring periods once patients are sufficiently awake and attentive within the ICU, at ICU discharge and again at acute hospital discharge. Measurements of patients muscle strength and physical function will also be made at the time of accelerometry.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ≥ 18 years of age
* Patient is/was intubated (endotracheal, nasotracheal or tracheostomy) and required ≥ 5 days of mechanical ventilation (irrespective of reason for ventilatory support)

Exclusion Criteria:

* Unable to ambulate independently (either with or without gait aids) at least 10 meters within the last 3 months
* Ordinarily unable to understand written and spoken English sufficient to provide consent (e.g. due to non-English speaking background or pre-existing cognitive impairment)
* Assessed by medical staff as approaching imminent death or withdrawal of medical management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU who are sufficiently awake and attentive (according to pre-determined awakening criteria) following at least 5 days of consecutive invasive mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Physical activity time | Change between events (each event assessed over 24 hours): From closest to the date of awakening in ICU (after at least 5 days of mechanical ventilation, assessed up to 4 months) to closest to the date of ICU discharge (assessed up to 6 months)
  Total time in minutes over 24 hours periods spent: at light, moderate and vigorous activity thresholds, in body positions of standing, walking and upright. Minute data derived from 2 accelerometers worn concurrently on each measurement occasion (wrist worn geneactiv for activity thresholds and thigh worn activpal for body postures)
Physical activity bouts | Change between events (each event assessed over 24 hours): From closest to the date of awakening in ICU (after at least 5 days of mechanical ventilation, assessed up to 4 months) to closest to the date of ICU discharge (assessed up to 6 months)
  Total number of bouts of physical activity over 24 hours periods spent: in light, moderate and vigorous activity thresholds, in body positions of standing, walking and upright. Data on number of bouts derived from 2 accelerometers worn concurrently on each measurement occasion (wrist worn geneactiv for activity thresholds and thigh worn activpal for body postures)
Sedentary time | Change between events (each event assessed over 24 hours): From closest to the date of awakening in ICU (after at least 5 days of mechanical ventilation, assessed up to 4 months) to closest to the date of ICU discharge (assessed up to 6 months)
  Total time in minutes over 24 hours periods spent: at a sedentary activity threshold, and in body positions of sitting/lying. Minute data derived from 2 accelerometers worn concurrently on each measurement occasion (wrist worn geneactiv for activity thresholds and thigh worn activpal for body postures)
Sedentary bouts | Change between events (each event assessed over 24 hours): From closest to the date of awakening in ICU (after at least 5 days of mechanical ventilation, assessed up to 4 months) to closest to the date of ICU discharge (assessed up to 6 months)
  Total number of bouts of sedentary time over 24 hours periods spent: at a sedentary activity threshold, and in body positions of sitting/lying. Data on number of bouts derived from 2 accelerometers worn concurrently on each measurement occasion (wrist worn geneactiv for activity thresholds and thigh worn activpal for body postures)
Physical activity time | Change between events (each event assessed over 24 hours): From closest to the date of awakening in ICU (after at least 5 days of mechanical ventilation, assessed up to 4 months) to closest to the date of hospital discharge (assessed up to 12 months)
  Total time in minutes over 24 hours periods spent: at light, moderate and vigorous activity thresholds, in body positions of standing, walking and upright. Minute data derived from 2 accelerometers worn concurrently on each measurement occasion (wrist worn geneactiv for activity thresholds and thigh worn activpal for body postures)
Physical activity bouts | Change between events (each event assessed over 24 hours): From closest to the date of awakening in ICU (after at least 5 days of mechanical ventilation, assessed up to 4 months) to closest to the date of hospital discharge (assessed up to 12 months)
  Total number of bouts of physical activity over 24 hours periods spent: in light, moderate and vigorous activity thresholds, in body positions of standing, walking and upright. Data on number of bouts derived from 2 accelerometers worn concurrently on each measurement occasion (wrist worn geneactiv for activity thresholds and thigh worn activpal for body postures)
Sedentary time | Change between events (each event assessed over 24 hours): From closest to the date of awakening in ICU (after at least 5 days of mechanical ventilation, assessed up to 4 months) to closest to the date of hospital discharge (assessed up to 12 months)
  Total time in minutes over 24 hours periods spent: at a sedentary activity threshold, and in body positions of sitting/lying. Minute data derived from 2 accelerometers worn concurrently on each measurement occasion (wrist worn geneactiv for activity thresholds and thigh worn activpal for body postures)
Sedentary bouts | Change between events (each event assessed over 24 hours): From closest to the date of awakening in ICU (after at least 5 days of mechanical ventilation, assessed up to 4 months) to closest to the date of hospital discharge (assessed up to 12 months)
  Total number of bouts of sedentary time over 24 hours periods spent: at a sedentary activity threshold, and in body positions of sitting/lying. Data on number of bouts derived from 2 accelerometers worn concurrently on each measurement occasion (wrist worn geneactiv for activity thresholds and thigh worn activpal for body postures)
Physical activity time | Change between events (each event assessed over 24 hours): From closest to the date of ICU discharge (assessed up to 6 months) to closest to the date of hospital discharge (assessed up to 12 months)
  Total time in minutes over 24 hours periods spent: at light, moderate and vigorous activity thresholds, in body positions of standing, walking and upright. Minute data derived from 2 accelerometers worn concurrently on each measurement occasion (wrist worn geneactiv for activity thresholds and thigh worn activpal for body postures)
Physical activity bouts | Change between events (each event assessed over 24 hours): From closest to the date of ICU discharge (assessed up to 6 months) to closest to the date of hospital discharge (assessed up to 12 months)
  Total number of bouts of physical activity over 24 hours periods spent: in light, moderate and vigorous activity thresholds, in body positions of standing, walking and upright. Data on number of bouts derived from 2 accelerometers worn concurrently on each measurement occasion (wrist worn geneactiv for activity thresholds and thigh worn activpal for body postures)
Sedentary time | Change between events (each event assessed over 24 hours): From closest to the date of ICU discharge (assessed up to 6 months) to closest to the date of hospital discharge (assessed up to 12 months)
  Total time in minutes over 24 hours periods spent: at a sedentary activity threshold, and in body positions of sitting/lying. Minute data derived from 2 accelerometers worn concurrently on each measurement occasion (wrist worn geneactiv for activity thresholds and thigh worn activpal for body postures)
Sedentary bouts | Change between events (each event assessed over 24 hours): From closest to the date of ICU discharge (assessed up to 6 months) to closest to the date of hospital discharge (assessed up to 12 months)
  Total number of bouts of sedentary time over 24 hours periods spent: at a sedentary activity threshold, and in body positions of sitting/lying. Data on number of bouts derived from 2 accelerometers worn concurrently on each measurement occasion (wrist worn geneactiv for activity thresholds and thigh worn activpal for body postures)

SECONDARY OUTCOMES:
Peripheral muscle strength | Change between events (each event assessed within 24 hours): From closest to the date of awakening in ICU (after at least 5 days of mechanical ventilation, assessed up to 4 months) to closest to the date of ICU discharge (assessed up to 6 months)
  Assessed with the medical research council (MRC) sum score, reported as a raw score /60 and categorically (yes/no) to indicate the presence of ICU acquired weakness (scores < 48/60 indicative of clinically significant weakness)
Peripheral muscle strength | Change between events (each event assessed within 24 hours): From closest to the date of awakening in ICU (after at least 5 days of mechanical ventilation, assessed up to 4 months) to closest to the date of hospital discharge (assessed up to 12 months)
  Assessed with the medical research council (MRC) sum score, reported as a raw score /60 and categorically (yes/no) to indicate the presence of ICU acquired weakness (scores < 48/60 indicative of clinically significant weakness)
Peripheral muscle strength | Change between events (each event assessed within 24 hours): From closest to the date of ICU discharge (assessed up to 6 months) to closest to the date of hospital discharge (assessed up to 12 months)
  Assessed with the medical research council (MRC) sum score, reported as a raw score /60 and categorically (yes/no) to indicate the presence of ICU acquired weakness (scores < 48/60 indicative of clinically significant weakness)
Hand grip strength | Change between events (each event assessed within 24 hours): From closest to the date of awakening in ICU (after at least 5 days of mechanical ventilation, assessed up to 4 months) to closest to the date of ICU discharge (assessed up to 6 months)
  Assessed with hand grip dynamometry in kilograms
Hand grip strength | Change between events (each event assessed within 24 hours): From closest to the date of awakening in ICU (after at least 5 days of mechanical ventilation, assessed up to 4 months) to closest to the date of hospital discharge (assessed up to 12 months)
  Assessed with hand grip dynamometry in kilograms
Hand grip strength | Change between events (each event assessed within 24 hours): From closest to the date of ICU discharge (assessed up to 6 months) to closest to the date of hospital discharge (assessed up to 12 months)
  Assessed with hand grip dynamometry in kilograms
Low level physical function/mobility | Change between events (each event assessed within 24 hours): From closest to the date of awakening in ICU (after at least 5 days of mechanical ventilation, assessed up to 4 months) to closest to the date of ICU discharge (assessed up to 6 months)
  Assessed with the PFIT (physical function in ICU test), reported as an interval score /10
Low level physical function/mobility | Change between events (each event assessed within 24 hours): From closest to the date of awakening in ICU (after at least 5 days of mechanical ventilation, assessed up to 4 months) to closest to the date of hospital discharge (assessed up to 12 months)
  Assessed with the PFIT (physical function in ICU test), reported as an interval score /10
Low level physical function/mobility | Change between events (each event assessed within 24 hours): From closest to the date of ICU discharge (assessed up to 6 months) to closest to the date of hospital discharge (assessed up to 12 months)
  Assessed with the PFIT (physical function in ICU test), reported as an interval score /10
High level physical function/mobility | Change between events (each event assessed within 24 hours): From closest to the date of awakening in ICU (after at least 5 days of mechanical ventilation, assessed up to 4 months) to closest to the date of ICU discharge (assessed up to 6 months)
  Assessed with the DEMMI (deMorton mobility index), reported as an interval score /100
High level physical function/mobility | Change between events (each event assessed within 24 hours): From closest to the date of awakening in ICU (after at least 5 days of mechanical ventilation, assessed up to 4 months) to closest to the date of hospital discharge (assessed up to 12 months)
  Assessed with the DEMMI (deMorton mobility index), reported as an interval score /100
High level physical function/mobility | Change between events (each event assessed within 24 hours): From closest to the date of ICU discharge (assessed up to 6 months) to closest to the date of hospital discharge (assessed up to 12 months)
  Assessed with the DEMMI (deMorton mobility index), reported as an interval score /100

OTHER OUTCOMES:
Intensive Care unit (ICU) length of stay | Time to event: from the date of hospital admission to the date of ICU discharge (up to 6 months)
  Based on hospital record data, reported in number of days. Associations with primary outcomes to be reported.
Acute hospital length of stay | Time to event: from the date of hospital admission to the date of hospital discharge (up to 12 months)
  Based on hospital record data, reported in number of days. Associations with primary outcomes to be reported.
Discharge destination | Event: date of hospital discharge (up to 12 months)
  Based on hospital record data, categorised as home, inpatient rehabilitation, another acute/community hospital, nursing home, other. Associations with primary outcomes to be reported.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baldwin CE, Rowlands AV, Fraysse F, Johnston KN. The sedentary behaviour and physical activity patterns of survivors of a critical illness over their acute hospitalisation: An observational study. Aust Crit Care. 2020 May;33(3):272-280. doi: 10.1016/j.aucc.2019.10.006. Epub 2019 Dec 6. PMID 31813736